CLINICAL TRIAL: NCT01924728
Title: A Randomized, Double-blind, Placebo Controlled Clinical Trial to Investigate the Effects of Transpelvic Magnetic Stimulation (Using QRS®-1010 PelviCenter) in Patients With Stress Urinary Incontinence.
Brief Title: Efficacy of Magnetic Stimulation for Stress Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: QRS Asia Sdn Bhd (Industry)
Collaborators: Universiti Sains Malaysia (Other); Island Hospital (Other); Penang Adventist Hospital (Unknown)
Responsible Party: Principal Investigator, Lim Renly, M. Pharm, QRS Asia Sdn Bhd
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: QRSPelvicenter
Record Dates: First submitted 2013-08-14; First posted 2013-08-16 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Magnetic stimulation (Active Comparator): Active magnetic stimulation delivered to the pelvic floor muscles
  Interventions: Device: Magnetic stimulation
- Sham magnetic stimulation (Sham Comparator): Sham magnetic stimulation delivered to the pelvic floor muscles
  Interventions: Device: Sham magnetic stimulation

INTERVENTIONS:
Device: Magnetic stimulation — 50Hz active magnetic stimulation (coil position 100%) delivered to the pelvic floor muscles
  Arms: Magnetic stimulation
Device: Sham magnetic stimulation — 50Hz sham magnetic stimulation (coil position 0%) delivered to the pelvic floor muscles
  Arms: Sham magnetic stimulation

SUMMARY:
The aim of the study is to investigate the effects of QRS®-1010 PelviCenter in female patients with stress urinary incontinence.

Based on the available data on magnetic stimulation, the investigators hypothesize that magnetic stimulation via QRS®-1010 PelviCenter will reduce the number and amount of urinary leakage upon exertion as well as improve patients' quality of life.

DETAILED DESCRIPTION:
A total of 120 female patients will be randomly assigned into two treatment groups (active arm and sham arm) in a 1:1 ratio. The standard QRS®-1010 PelviCenter treatment plan involves 16 sessions of 20 minutes each. Each subject will attend 2 sessions per week (total 16 sessions).

ELIGIBILITY:
Inclusion Criteria:

* Female aged at least 21 years old
* Demonstration of stress urinary incontinence by vaginal examination with half full bladder (200 to 250ml)
* ICIQ UI SF score ≥ 6 points
* Able and agree to carry out one hour pad test

Exclusion Criteria:

* Acute severe infections
* Urinary tract infections and hematuria, active vaginal lesions or infections
* Pelvic organ prolapse stage III and IV, severe urethral sphincter weakness/defect, suspected fistula
* Severe cardiac arrhythmia
* Cardiac pacemaker or other implanted metallic devices
* History of pelvic irradiation
* Pregnant, or actively trying to conceive.
* Neurologic conditions such as epilepsy, Parkinson disease, multiple sclerosis
* Patient who has been treated with electromagnetic stimulation
* Concurrent medications with alpha-adrenergic antagonists (e.g. terazosin, tamsulosin, doxazosin), diuretics, serotonin/norepinephrine reuptake inhibitors (SNRIs) or any other medications known to worsen incontinence.
* Post void residual volume of ≥ 200ml
* Random blood sugar >10 mmol/L
* Patient who had pelvic or gynaecological surgery for less than three weeks
* Patient scheduled for pelvic or gynaecological surgery in the next eight weeks

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-09; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change in International consultation on incontinence questionnaire for urinary incontinence-short form (ICIQ-UI SF) | Baseline, Week 4, 8. Follow-up at 3-,6- and 12-months post treatment

SECONDARY OUTCOMES:
Change in Incontinence Episode Frequency (IEF) | Baseline, Week 4, 8. Follow-up at 3-,6- and 12-months post treatment
Change in 1-hour exercise (stress) pad test | Baseline, Week 4, 8. Follow-up at 3-,6- and 12-months post treatment
Change in Patient Global Impression of Improvement (PGI-I) | Week 4, 8. Follow-up at 3-,6- and 12-months post treatment
Change in International consultation on incontinence questionnaire-Lower Urinary Tract Symptoms Quality of Life (ICIQ-LUTSqol) | Baseline, Week 4, 8. Follow-up at 3-,6- and 12-months post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Liong Men Long, MBBS, Principal Investigator — Island Hospital, Penang
Locations (1):
- Island Hospital, George Town, Pulau Pinang, Malaysia

REFERENCES:
- [Derived] Lim R, Liong ML, Leong WS, Khan NA, Yuen KH. Magnetic stimulation for stress urinary incontinence: study protocol for a randomized controlled trial. Trials. 2015 Jun 21;16:279. doi: 10.1186/s13063-015-0803-1. PMID 26093910